CLINICAL TRIAL: NCT04513847
Title: PsoVac: A Psoriatic Patient-based Survey on the Understanding of the Use of Vaccines While on Biologics During the Covid-19 Pandemic
Brief Title: PsoVac: Educational Needs re Vaccines for Biologic Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: Dermatrials Research (Other)
Responsible Party: Principal Investigator, Ronald Vender MD FRCPC, Associate Clinical Professor, Division of Dermatology MD FRCPC, Dermatrials Research
Other Study IDs: Pso-Vac
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Psoriasis; Covid19
Keywords: Education; Vaccine; Biologic
MeSH Terms: conditions — Psoriasis; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Psoriasis patients treated with non-biologic
- Non-Control: Psoriasis patients treated with biologic

SUMMARY:
To determine if there is a need for further education on vaccines with psoriasis patients who are on a biologic. In regards to the COVID-19, it is important that psoriasis patients - whether on a biologic or not - understand whether they can have certain vaccines. That will depend on the type of vaccine that becomes available.

ELIGIBILITY:
Inclusion Criteria:

* psoriasis patient

Exclusion Criteria:

* no exclusions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dermatology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 661 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients not understanding the interaction of vaccines and their biologic, assessed with voluntary survey. | Data will be collected over a span of 3 months
  Assessment is based upon survey responses. By answering multiple questions we will determine if more education is needed based on the answers.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatrials Research, Hamilton, Ontario, Canada